CLINICAL TRIAL: NCT01195103
Title: A Prospective Randomized Study to Assess the Efficacy and Safety of Bolus-dose Lusedra (Fospropofol Disodium) 6.5 mg/kg or 10 mg/kg Versus a Placebo (With Midazolam Rescue) for Minimal-to-moderate Sedation in Patients Undergoing Procedural Sedation for Regional Anesthesia Blocks Prior to Orthopedic Surgery
Brief Title: Lusedra (Fospropofol Disodium) for Minimal to Moderate Sedation for Regional Anesthesia Block Prior to Orthopedic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding terminated by funding source.
Sponsor: Mayo Clinic (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: John B Leslie MD MBA, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-000721
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Procedural Sedation; Regional Anesthesia Block; Orthopedic Surgery
Keywords: Procedural sedation; Regional Anesthesia block; Orthopedic surgery; Lusedra; Fospropofol disodium; Midazolam
MeSH Terms: interventions — fospropofol; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 mg/kg Lusedra (Experimental): 10 mg/kg Lusedra initial bolus.
  Interventions: Drug: Fospropofol disodium; Drug: Fentanyl
- 6.5 mg/kg Lusedra (Active Comparator): 6.5 mg/kg Lusedra initial bolus.
  Interventions: Drug: Fospropofol disodium; Drug: Fentanyl
- Placebo + Midazolam (Active Comparator): Placebo initial bolus with dose of midazolam based on patient's weight
  Interventions: Drug: Placebo + Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Fospropofol disodium — 10 mg/kg bolus
  Other Names: Lusedra
  Arms: 10 mg/kg Lusedra
Drug: Fospropofol disodium — 6.5 mg/kg bolus
  Other Names: Lusedra
  Arms: 6.5 mg/kg Lusedra
Drug: Placebo + Midazolam — Placebo bolus plus midazolam. The dose of midazolam will be based on the patient's weight: 1 mg for patients <60 kg; 1.5 mg for patients ≥60 kg to <90 kg; or 2 mg for patients ≥90 kg
  Other Names: Versed
  Arms: Placebo + Midazolam
Drug: Fentanyl — All patients will receive a single dose of IV fentanyl (approximately 1 μg/kg not to exceed: 50 μg for patients <60 kg; 75 μg for patients ≥90 kg) five minutes prior to the initial dose of sedative.
  Other Names: Fentanyl Citrate; Sublimaze

SUMMARY:
How does Lusedra compare with current standard of care (midazolam) for minimal to moderate sedation for regional anesthesia blocks prior to orthopedic surgery?

DETAILED DESCRIPTION:
The study overall is aimed at establishing the superiority of a single intravenous bolus-dose of Lusedra for routine use in preoperative regional blocks that avoids deeper levels of sedation and increased risk of nerve damage in an over-sedated individual. The shorter half-life of Lusedra should also demonstrate a superior recovery profile compared to midazolam when used as a rescue comparator. While this study will only enroll patients undergoing regional blocks prior to orthopedic surgery, the clinical utility and value of the larger initial intravenous dosing for Lusedra may be evident for many different monitored anesthesia care anesthetic management situations requiring rapid and effective onset of effects.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective orthopedic surgery
* With a regional block prior to surgery
* Able to consent and complete the assessments and procedures
* If female, must be surgically sterile, postmenopausal, or not pregnant or lactating and using an acceptable method of birth control for at least 1 month prior to surgery with a negative urine pregnancy test at screening
* American Society of Anesthesiologists Physical Classification System status category P1 to P4

Exclusion Criteria:

* History of allergic reaction or hypersensitivity to any anesthetic agent, opioid, or benzodiazepine
* Fentanyl citrate injection or midazolam hydrocholoride injection contraindicated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Leslie, MD MBA, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Mayo Clinic, Arizona from March 1 - 11, 2011.
Period: Overall Study
Arm/Group | 10 mg/kg Lusedra | 6.5 mg/kg Lusedra | Placebo + Midazolam
Started | 6 | 2 | 5
Completed | 5 (One patient withdrew after randomization but before received study drug.) | 2 | 5
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg/kg Lusedra | 6.5 mg/kg Lusedra | Placebo + Midazolam | Total
Number analyzed (Participants) | 6 | 2 | 5 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 73.2 (7.0) | 71.5 (4.3) | 72 (12) | 72.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4 | 8
  Male | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sedation Within 4 Minutes
Description: Percentage of patients achieving a Modified Observer's Assessment of Alertness/Sedation Scale score less than or equal to 4, and the block procedure initiated, within 4 minutes of the administration of the first bolus of study drug. The Modified Observer's Assessment of Alertness/Sedation Scale ranges from 0 (does not respond to deep stimulus) to 6 (agitated). The score of 4 equals "lethargic response to name spoken in normal tone."
Time Frame: approximately 4 minutes after administration of first bolus of study drug
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg/kg Lusedra | 6.5 mg/kg Lusedra | Placebo + Midazolam
Number analyzed (Participants) | 5 | 2 | 5
percentage of participants | 100 | 50 | 40

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from the time of drug administration until entry into the operating room. Patients were sedated again for the surgery. We only studied the first sedation.
Description: No adverse event data were collected for the patient who withdrew prior to receiving study drug, so that patient was not included in the assessment of adverse events.
Arm/Group | 10 mg/kg Lusedra | 6.5 mg/kg Lusedra | Placebo + Midazolam
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 1/2 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/kg Lusedra (N=5) | 6.5 mg/kg Lusedra (N=2) | Placebo + Midazolam (N=5)
apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/kg Lusedra (N=5) | 6.5 mg/kg Lusedra (N=2) | Placebo + Midazolam (N=5)
deep sedation (Nervous system disorders) | 5 (5) | 0 (0) | 1 (1)
delayed recovery from sedation (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
puritis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early because funding was terminated by the funding source.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No